CLINICAL TRIAL: NCT02722330
Title: Evaluation of Audiological Outcomes and Subjective Benefits of Cochlear Baha® 5 SuperPower Sound Processor on the Baha® Attract™ System
Brief Title: Evaluation of Cochlear Baha 5 SuperPower Sound Processor on the Baha Attract System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear Bone Anchored Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CBAS5619
Record Dates: First submitted 2016-02-17; First posted 2016-03-30 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Single Sided Sensorineural Deafness; Mixed Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baha 5 SuperPower on Baha Attract System (Experimental): The device involves the following parts:
  The sound processor unit, an actuator unit and a cable, the Sound Processor Magnet (SP Magnet) of the Baha Attract System, the BIM400 Baha Implant Magnet that is fixated to the BI300 Implant, a snap coupling.
  Interventions: Device: Baha 5 SuperPower on Baha Attract System

INTERVENTIONS:
Device: Baha 5 SuperPower on Baha Attract System — The Investigational device involves the following parts: the sound processor unit, an actuator unit and a cable that connects the sound processor and actuator units. The actuator unit is attached to the Sound Processor Magnet (SP Magnet) of the Baha Attract System which is pulled towards the BIM400 Baha Implant Magnet that is fixated to the BI300 Implant. The actuator unit can also be connected to the Baha Softband via a snap coupling.

SUMMARY:
The aim of this clinical investigation is to evaluate objective and subjective hearing performance with the Cochlear Baha 5 SuperPower Sound Processor on the Baha Attract System, compared to the unaided hearing performance. Comparison of audiological test results with the same sound processor on a Baha Softband will also be performed. Short term safety parameters will be collected.

DETAILED DESCRIPTION:
The Cochlear Baha bone conduction hearing implant offers two alternative ways to transmit vibrations from the external sound processor to the osseointegrated implant: The Baha Connect System uses a skin-penetrating abutment and allows direct bone conduction. The Baha Attract System uses a magnetic connection through intact skin. Magnetic bone conduction hearing implants have the advantage over skin-penetrating systems of eliminating the daily cleaning of the site and are perceived as a more cosmetically appealing by some subjects. With modern sound processor technology, it is possible to obtain good sound transmission despite the soft tissue attenuation that is inherent to magnetic bone conduction hearing implants. Clinical investigations have shown that the Baha Attract System, when used in combination with existing head-worn sound processors within the Premium (e.g. BP100, Baha 4 Sound Processors) and Power (BP110 Sound processor) segments, provides good hearing outcomes in subjects with conductive and mild mixed hearing loss.

The Cochlear Baha 5 SuperPower Sound Processor is the first head-worn sound processor within the Super Power segment and has a fitting range of 65 dBHL. It is CE marked and is intended for subjects with mixed hearing loss or single-sided sensorineural deafness (SSD). It can be used with the Baha Connect and Baha Attract Systems and with a Baha Softband. When used in combination with the Baha Attract System, it will be able to compensate for a larger sensorineural component than the current Premium and Power sound processors and, hence, will allow more subjects to benefit from the Baha Attract System. The combination Baha Attract System with Baha 5 SuperPower Sound Processor is the most powerful non-skin penetrating bone conduction hearing implant solution available today.

The Baha 5 SuperPower Sound Processor includes discreet design, advanced signal processing and improved connectivity to external sound sources. The new sound processor supports Cochlear's 2.4 GHz wireless protocol and is programmable with a new version of the Baha 5 Fitting Software.

The aim of this clinical investigation is to evaluate objective and subjective hearing performance with the Cochlear Baha 5 SuperPower Sound Processor on the Baha Attract System, compared to the unaided hearing performance. Comparison of audiological test results with the same sound processor on a Baha Softband will also be performed. Short term safety parameters will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 18 years of age
* Mixed hearing loss in the ear to be implanted. Bone conduction thresholds with pure tone average (PTA4, Mean of 0.5, 1, 2 and 4kHz) of 30-55 dBHL or
* Single-sided sensorineural deafness: Bone conduction thresholds with a pure tone average [PTA4, Mean of 0.5, 1, 2 and 4 kHz] of lower or 30 dBHL in the best ear. Subjects who have, for some reason, experienced no or limited benefit from other sound processors when tested on a Baha Softband.
* Subjects suitable for surgery according to the recommended surgical procedure for Cochlear Baha 5 SuperPower with no previous implant on the side to be investigated.
* Signed inform consent.

Exclusion Criteria:

* Subject scheduled for simultaneous bilateral implant surgery. The investigation is limited to subjects with unilateral use of the Investigational device (however, bilateral hearing loss is not an exclusion criterion).
* Suitable implant position for the BI300 Implant (4 mm or 3 mm) not found during surgery due to insufficient bone quality and/or bone thickness
* Less than 3 mm soft tissue thickness at the planned implant site. (Intra-operative exclusion criteria judged by the surgeon at Visit 1 or Visit 2 according to local practice).
* Subjects that have received radiation therapy at the same side of the skull where the Investigational device will be positioned.
* Uncontrolled diabetes as judged by the investigator.
* Condition that could jeopardise osseointegration and/or wound healing (e.g. osteoporosis, psoriasis and long-term systemic use of corticosteroids) or condition that may have an impact on the outcome of the investigation as judged by the investigator.
* Unable to follow investigational procedures, e.g. to complete quality of life scales.
* Participation in another clinical investigation with pharmaceutical and/or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaydip Ray, Professor, Principal Investigator — Royal Hallamshire Hospital; César Orús, Dr, Principal Investigator — Hospital de Sant Pau; Paul Van de Heyning, Professor, Principal Investigator — University Hospital, Antwerp; Jesper Schmidt, Dr, Principal Investigator — Odense University Hospital
Locations (4):
- Antwerp University Hospital, Antwerp, Belgium
- Odense University Hospital, Odense, Denmark
- Hospital de Sant Pau, Barcelona, Spain
- Royal Hallamshire Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Baha 5 SuperPower on Baha Attract System: The device involves the following parts:
  The sound processor unit, an actuator unit and a cable, the Sound Processor Magnet (SP Magnet) of the Baha Attract System, the BIM400 Baha Implant Magnet that is fixated to the BI300 Implant, a snap coupling.
  Baha 5 SuperPower on Baha Attract System: The Investigational device involves the following parts: the sound processor unit, an actuator unit and a cable that connects the sound processor and actuator units. The actuator unit is attached to the Sound Processor Magnet (SP Magnet) of the Baha Attract System which is pulled towards the BIM400 Baha Implant Magnet that is fixated to the BI300 Implant. The actuator unit can also be connected to the Baha Softband via a snap coupling.
Period: Overall Study
Arm/Group | Baha 5 SuperPower on Baha Attract System
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 10
  Denmark | 2
  United Kingdom | 6
  Spain | 5
Type of hearing loss in treatment ear [Count of Participants; unit: Participants]
  Mixed hearing loss | 23
  Single-sided sensorineural deafness | 0
Treatmen ear [Count of Participants; unit: Participants]
  Right | 13
  Left | 10
Does the subject use a hearing aid in the treament ear [Count of Participants; unit: Participants]
  Yes | 10
  No | 13
Does the subject use a hearing aid in the non-treament ear [Count of Participants; unit: Participants]
  Yes | 9
  No | 14

OUTCOME MEASURES:

1. Primary Outcome: Audiometry; Free Field Thresholds. Pure Tone Average PTA4,Unaided vs Aided
Description: Change of hearing performance PTA4 [Mean of 0.5, 1, 2 and 4 kHz] from the unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL | -27.7 (9.0)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

2. Secondary Outcome: Change of the Self-reported Assessments of Hearing Outcome Using Abbreviated Profile of Hearing Aid Benefit (APHAB) From the Unaided Hearing Situation at Pre-operation With the Investigational Device on the Attract System, at 12 Weeks.
Description: The APHAB is a 24-item self-assessment questionnaire evaluating the benefit experienced by the subject when using hearing amplification compared to the unaided situation. It comprises of four subscales: Ease of Communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV). The Global score is the mean of the subscales. All subscales are scored in the same way.
  The scores show how frequently (%) clients experience performance problems and varies between 0-100, 0 indicates no problems, 100 indicates always problem. Benefit is then calculated by subtracting the aided average from the unaided average. The theoretical benefit score could vary between -100 to + 100. The higher the score the better benefit and positive score indicates an improvement, a negative value an impairment.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
score on a scale
  Ease of communication | 44.8 (33.1)
  Reverberation | 31.5 (23.8)
  Background noise | 37.7 (25.1)
  Aversiveness | -16.6 (27.3)
  Global score | 38.0 (24.2)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Ease of communication; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; Reverberation; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed rank Test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; Background noise; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed rank Test
Statistical Analysis 4: Comparison: Baha 5 SuperPower on Baha Attract System; Aversiveness; Test type: Superiority or Other; p = 0.0004, Wilcoxon Signed rank Test
Statistical Analysis 5: Comparison: Baha 5 SuperPower on Baha Attract System; Global score; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed rank Test

3. Secondary Outcome: Change of the Self-reported Assessments of Hearing Outcome Using Speech, Spatial and Qualities of Hearing Scale (SSQ-12) From the Unaided Hearing Situation at Pre-operation With the Investigational Device on the Attract System, Aided at 12 Weeks.
Description: The SSQ-12 is comprised of 12 items using the response format on a scale from 0 to 10, were 0 equals no ability and 10 equals perfect ability. These are divided into three sub-scales and the questions 1-5 are from the speech sub-scale, 6-8 from the spatial, and 9-12 from the qualities sub-scale. The three sub-scales are the average of the questions within. A 'not applicable' option is given for each item.
  The change from unaided to aided hearing is then calculated and the theoretical score could vary between -10 to + 10. The higher the score the better benefit and positive score indicates improved hearing, a negative value an impaired hearing.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
score on a scale
  Speech scale | 3.59 (1.9)
  Spatial scale | 2.37 (2.08)
  Qualities scale | 3.51 (2.16)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Speech scale; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; Spatial scale; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; Qualities scale; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

4. Secondary Outcome: Audiometry; Free Field Thresholds. Pure Tone Average PTA4 Unaided vs Aided
Description: Change of hearing performance PTA4 [Mean of 0.5, 1, 2 and 4 kHz] from the unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL | -27.0 (9.7)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

5. Secondary Outcome: Audiometry; Free Field Thresholds Per Frequency, Unaided vs Aided
Description: Change of hearing performance free field tresholds per frequency [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 kHz] from unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL
  250 Hz | -20.7 (13.3)
  500 Hz | -27.6 (11.8)
  750 Hz | -33.0 (13.5)
  1000 Hz | -31.5 (11.0)
  1500 Hz | -35.9 (11.1)
  2000 Hz | -30.0 (10.9)
  3000Hz | -20.9 (16.1)
  4000 Hz | -18.9 (16.0)
  6000 Hz | -19.5 (13.9)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; 250 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; 500 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; 750 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Baha 5 SuperPower on Baha Attract System; 1000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Baha 5 SuperPower on Baha Attract System; 1500 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Baha 5 SuperPower on Baha Attract System; 2000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Baha 5 SuperPower on Baha Attract System; 3000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Baha 5 SuperPower on Baha Attract System; 4000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 9: Comparison: Baha 5 SuperPower on Baha Attract System; 6000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

6. Secondary Outcome: Audiometry; Free Field Thresholds Per Frequency, Unaided vs Aided
Description: Change of hearing performance free field tresholds per frequency [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 kHz] from unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL
  250 Hz | -24.3 (11.3)
  500 Hz | -27.6 (12.0)
  750 Hz | -33.0 (13.8)
  1000 Hz | -32.2 (11.2)
  1500 Hz | -35.9 (11.1)
  2000 Hz | -32.4 (10.1)
  3000 Hz | -23.9 (12.3)
  4000 Hz | -18.5 (13.7)
  6000 Hz | -23.4 (14.8)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; 250 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; 500 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; 750 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Baha 5 SuperPower on Baha Attract System; 1000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Baha 5 SuperPower on Baha Attract System; 1500 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Baha 5 SuperPower on Baha Attract System; 2000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Baha 5 SuperPower on Baha Attract System; 3000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Baha 5 SuperPower on Baha Attract System; 4000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 9: Comparison: Baha 5 SuperPower on Baha Attract System; 6000 Hz; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

7. Secondary Outcome: Free Field; - Adaptive Speech Recognition in Noise, Unaided vs Aided
Description: Change of hearing performance free field - adaptive speech recognition in noise from unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 17
dB | -8.56 (6.22)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p = 0.002, Wilcoxon Signed Rank test

8. Secondary Outcome: Free Field; - Adaptive Speech Recognition in Noise, Unaided vs Aided
Description: Change of hearing performance free field - adaptive speech recognition in noise from unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 17
dB | -8.41 (5.13)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p = 0.0024, Wilcoxon Signed Rank test

9. Secondary Outcome: Free Field; - Speech Recognition in Quiet, Unaided vs Aided
Description: Change of hearing performance free field - speech recognition in quiet from the unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage (%) correct words
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Percentage (%) correct words
  Speech Presentation Level 50 dB | 34.1 (31.4)
  Speech Presentation Level 65 dB | 43.3 (27.6)
  Speech Presentation Level 80 dB | 34.5 (33.1)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Speech Presentation Level 50 dB; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; Speech Presentation Level 65 dB; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; Speech Presentation Level 80 dB; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

10. Secondary Outcome: Free Field; - Speech Recognition in Quiet, Unaided vs Aided
Description: Change of hearing performance free field - speech recognition in quiet from the unaided hearing situation at pre-operation with the Investigational device on the attract system, aided at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage (%) correct words
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Percentage (%) correct words
  Speech Presentation Level 50 dB | 35.7 (29.6)
  Speech Presentation Level 65 dB | 49.0 (29.5)
  Speech Presentation Level 80 dB | 39.2 (32.9)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Speech Presentation Level 50 dB; Test type: Superiority or Other; p < 0.0001, Wolcoxon Signed rank test — All variable had the same p value (<0.0001)
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; Speech Presentation Level 65 dB; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; Speech Presentation Level 80 dB; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank test

11. Secondary Outcome: Audiometry; Free Field Thresholds. Pure Tone Average PTA4, Investigational Device vs Softband
Description: Change of hearing performance PTA4 [Mean of 0.5, 1, 2 and 4 kHz] from the situation with the same sound processor on a Baha soft band at pre-operation with the Investigational device on the attract system at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL | 2.55 (5.87)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p = 0.036, Wilcoxon Signed Rank test

12. Secondary Outcome: Audiometry; Free Field Thresholds. Pure Tone Average PTA4 [Mean of 0.5, 1, 2 and 4 kHz], Investigational Device vs Softband
Description: Change of hearing performance PTA4 from the situation with the same sound processor on a Baha soft band at pre-operation with the Investigational device on the attract system at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL | 1.9 (4.31)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p = 0.065, Wilcoxon Signed Rank test

13. Secondary Outcome: Audiometry; Free Field Thresholds Per Frequency, Investigational Device vs Softband
Description: Change of hearing performance free field tresholds per frequency [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 kHz] from the situation with same sound processor on a Baha softband with the Investigational device on the attract system at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL
  250 Hz | 1.3 (7.42)
  500 Hz | -2.61 (7.52)
  750 Hz | 1.09 (7.38)
  1000 Hz | 3.04 (6.70)
  1500 Hz | 1.52 (6.47)
  2000 Hz | 4.57 (8.25)
  3000 Hz | 5.65 (10.90)
  4000 Hz | 5.22 (12.29)
  6000 Hz | 7.62 (11.47)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; 250 Hz; Test type: Superiority or Other; p = 0.47, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; 500 Hz; Test type: Superiority or Other; p = 0.16, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; 750 Hz; Test type: Superiority or Other; p = 0.59, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Baha 5 SuperPower on Baha Attract System; 1000 Hz; Test type: Superiority or Other; p = 0.034, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Baha 5 SuperPower on Baha Attract System; 1500 Hz; Test type: Superiority or Other; p = 0.25, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Baha 5 SuperPower on Baha Attract System; 2000 Hz; Test type: Superiority or Other; p = 0.023, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Baha 5 SuperPower on Baha Attract System; 3000 Hz; Test type: Superiority or Other; p = 0.028, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Baha 5 SuperPower on Baha Attract System; 4000 Hz; Test type: Superiority or Other; p = 0.0075, Wilcoxon Signed Rank test
Statistical Analysis 9: Comparison: Baha 5 SuperPower on Baha Attract System; 6000 Hz; Test type: Superiority or Other; p = 0.0035, Wilcoxon Signed Rank test

14. Secondary Outcome: Audiometry; Free Field Thresholds Per Frequency, Investigational Device vs Softband
Description: Change of hearing performance free field tresholds per frequency [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 kHz] from the same sound processor on a Baha softband with the Investigational device on the attract system at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB HL
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
dB HL
  250 Hz | -2.39 (7.52)
  500 Hz | -2.61 (6.01)
  750 Hz | 1.09 (6.21)
  1000 Hz | 2.39 (6.89)
  1500 Hz | 1.52 (7.30)
  2000 Hz | 2.17 (6.54)
  3000 Hz | 2.61 (11.66)
  4000 Hz | 5.65 (10.69)
  6000 Hz | 2.50 (18.31)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; 250 Hz; Test type: Superiority or Other; p = 0.12, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; 500 Hz; Test type: Superiority or Other; p = 0.072, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; 750 Hz; Test type: Superiority or Other; p = 0.56, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Baha 5 SuperPower on Baha Attract System; 1000 Hz; Test type: Superiority or Other; p = 0.16, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Baha 5 SuperPower on Baha Attract System; 1500 Hz; Test type: Superiority or Other; p = 0.39, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Baha 5 SuperPower on Baha Attract System; 2000 Hz; Test type: Superiority or Other; p = 0.11, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Baha 5 SuperPower on Baha Attract System; 3000 Hz; Test type: Superiority or Other; p = 0.38, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Baha 5 SuperPower on Baha Attract System; 4000 Hz; Test type: Superiority or Other; p = 0.014, Wilcoxon Signed Rank test
Statistical Analysis 9: Comparison: Baha 5 SuperPower on Baha Attract System; 6000 Hz; Test type: Superiority or Other; p = 0.71, Wilcoxon Signed Rank test

15. Secondary Outcome: Free Field - Adaptive Speech Recognition in Noise, Investigational Device vs Softband
Description: Change of hearing performance free field - adaptive speech recognition in noise from the situation with the same sound processor on a Baha softband at pre-operation with the Investigational device on the attract system at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 17
dB | 1.19 (4.45)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p = 0.48, Wilcoxon Signed Rank test

16. Secondary Outcome: Free Field - Adaptive Speech Recognition in Noise, Investigational Device vs Softband
Description: Change of hearing performance free field - adaptive speech recognition in noise from the situation with the same sound processor on a Baha softband at pre-operation with the Investigational device on the attract system at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 17
dB | 1.42 (3.27)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; Test type: Superiority or Other; p = 0.11, Wilcoxon Signed Rank test

17. Secondary Outcome: Free Field - Speech Recognition in Quiet, Investigational Device vs Softband
Description: Change of hearing performance free field - speech recognition in quiet from the situation with the same sound processor on a Baha Softband with the Investigational device on the attract system at 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage (%) correct words
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Percentage (%) correct words
  Speech Presentation Level 50 dB | -10.5 (25.7)
  Speech Presentation Level 65 dB | -6.78 (18.37)
  Speech Presentation Level 80 dB | -1.86 (17.39)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; SPL 50 dB; Test type: Superiority or Other; p = 0.017, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; SPL 65 dB; Test type: Superiority or Other; p = 0.095, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; SPL 80 dB; Test type: Superiority or Other; p = 0.57, Wilcoxon Signed Rank test

18. Secondary Outcome: Free Field - Speech Recognition in Quiet, Investigational Device vs Softband
Description: Change of hearing performance free field - speech recognition in quiet from the situation with the same sound processor on a Baha Softband with the Investigational device on the attract system at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 17
dB
  Speech Presentation Level 50 dB | -9.00 (19.80)
  Speech Presentation Level 65 dB | -1.17 (16.52)
  Speech Presentation Level 80 dB | 2.82 (18.11)
Statistical Analysis 1: Comparison: Baha 5 SuperPower on Baha Attract System; SPL 50 dB; Test type: Superiority or Other; p = 0.096, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Baha 5 SuperPower on Baha Attract System; SPL 65 dB; Test type: Superiority or Other; p = 1.00, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Baha 5 SuperPower on Baha Attract System; SPL 80 dB; Test type: Superiority or Other; p = 0.41, Wilcoxon Signed Rank test

19. Secondary Outcome: Sound Processor Magnet Selection at 4 Weeks
Description: Information about sound processor magnet selection, type of SP magnet
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Participants
  SPM1 | 0
  SPM2 | 2
  SPM3 | 3
  SPM4 | 11
  SPM5 | 5
  SPM6 | 2

20. Secondary Outcome: Sound Processor Magnet Selection at 6 Weeks
Description: Information about sound processor magnet selection, type of SP magnet
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Participants
  SPM1 | 0
  SPM2 | 5
  SPM3 | 8
  SPM4 | 7
  SPM5 | 2
  SPM6 | 1

21. Secondary Outcome: Sound Processor Magnet Selection at 12 Weeks
Description: Information about sound processor magnet selection, type of SP magnet
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
Participants
  SPM1 | 2
  SPM2 | 3
  SPM3 | 8
  SPM4 | 10
  SPM5 | 0
  SPM6 | 0

22. Secondary Outcome: Daily Use of Sound Processor (Average Daily Use During the Last Week)
Description: Average daily use (hours/day) of the sound processor during the last week of the study
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
hours/day | 9.39 (3.54)

23. Other Pre Specified Outcome: Number of Adverse Events Related to the Treatment
Description: Number of adverse events related to the treatment during the 12 weeks treatment period
Time Frame: 12 weeks
Measure: Number; unit: events
Arm/Group | Baha 5 SuperPower on Baha Attract System
Number analyzed (Participants) | 23
events | 3

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Baha 5 SuperPower on Baha Attract System
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baha 5 SuperPower on Baha Attract System (N=23)
Pain/discomfort (General disorders) | 1 (2)
Other (Renal and urinary disorders) | 1 (1)
Presssure related skin complications (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days